CLINICAL TRIAL: NCT00904592
Title: A Study on TCM Comprehensive Protocol of Prevention and Control in Diabetic Retinopathy
Brief Title: A Study on Traditional Chinese Medicine (TCM) Comprehensive Protocol of Prevention and Control in Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2006BAI04A0401
Record Dates: First submitted 2008-12-24; First posted 2009-05-19 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; traditional chinese medicine
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qi ming granula (Experimental): Study group(combined therapy with Intervention of TCM): Basic therapy ＆ treating both on deficiency and stasis of blood.
  1. Therapy for DM: To control blood glucose, blood pressure, and serum lipid through drug, dietary management, exercise and education.
  2. Qi ming granula, Usage: 4.5g，po，tid.
  Interventions: Drug: Qi ming granula
- placebo comparator (Placebo Comparator): Control group: Basic therapy ＆ placebo
  1. Therapy for DM: To control blood glucose, blood pressure, and serum lipid through drug, dietary management , exercise and education.
  2. placebo,Usage: 4.5g，po，tid
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Qi ming granula — Qi ming granula Usage:4.5g，po，tid. duration:12 months/ arise Endpoint Event
  Other Names: QM
  Arms: Qi ming granula
Drug: Placebo Comparator — Control group: Basic therapy ＆ placebo
  1. Therapy for DM: To control blood glucose, blood pressure, and serum lipid through drug, dietary management , exercise and education.
  2. placebo,Usage: 4.5g，po，tid
  Other Names: PC
  Arms: placebo comparator

SUMMARY:
1. Title: A Study on TCM comprehensive protocol of Prevention and Control in Diabetic Retinopathy.
2. Objectives of study: To evaluate the Intervention effect of integrate control protocol on reducing the incidence rate of proliferative diabetic retinopathy, PRP and MVL. Then produce a high performance, optimize, convenient, applicable and demonstrated protocol of integrate control with Intervention of TCM and west medicine.
3. Study Type: Interventional
4. Study Design: Multi-center, Randomized, Blind (Subject, Investigator, Outcomes Assessor), Parallel Assignment, Positive controlled clinical study.
5. Sample size: 480 subjects , divided into test and control groups equally.
6. Primary endpoint: incidence rate of proliferative diabetic retinopathy, panretinal photocoagulation

DETAILED DESCRIPTION:
1. Primary outcome:

   * proliferative diabetic retinopathy
   * panretinal photocoagulation
2. Secondary outcome:

   * Vision, Funduscopy, Fundus photograph
   * Fundus fluorescein angiography
   * Visual Electrophysiology:FERG、OPs、PVEP.
   * Optical coherence tomography.
   * Symptoms scores of TCM.
   * The M0S short-form-36 heaIth survey(SF-36).
   * Visual Function Questionnaire-25(VFQ-25).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus.
* Diagnosed with non-proliferative diabetic retinopathy, including moderate and severe diabetic retinopathy
* and corrected VA≥45 letters(ETDRS), equivalent the decimal value of 0.16(20/125).
* Diagnosed with the syndrome and signs of TCM.
* HbA1C≤8.0%.
* Ages ranged from 35 to 75 years.
* Joined in the test voluntarily and signed the Informed consent by GCP regulation.

Exclusion Criteria:

* Complicating severe vitreous hemorrhage, or requiring laser and vitrectomy treatment.
* The patients who have been received the therapy of Retina laser photocoagulation.
* The patients whose dioptric media is so turbid that hard to evaluate the fundus picture.
* DMKA or other acute metabolic disturbance, or complicating severe acute infection within a month.
* Combined with other severe Diabetic complication.
* Having any allergic reaction to some drugs, food and pollen etc. or hypersensitiveness
* Pregnant or breast feeding.
* combined with primarily severe diseases such as cardiovascular, hepatic，renal illness ,hemopoietic system disease, and psychosis.
* Combined with glaucoma, uveitis, ocular neuropathy and severe cataract etc.
* Participated in other clinical trial within 3 month.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2008-09; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
incidence rate of proliferative diabetic retinopathy, panretinal photocoagulation | 12 months

SECONDARY OUTCOMES:
Symptoms scores of TCM | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junguo Duan, Principal Investigator — Chengdu University of TCM
Locations (1):
- Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19802544?itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_RVDocSum&ordinalpos=1